CLINICAL TRIAL: NCT06267040
Title: Linguistic and Clinical Validation of the Arabic Version of Acute Cystitis Symptom Score (ACCS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Kindy College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 17 Al-KindyCM
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-01

CONDITIONS: Cystitis Acute
Keywords: uncomplicated cystitis; linguistic validation; Acute Cystitis symptom score; ACSS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women diagnosed with uncomplicated cystitis: women older than 18 years diagnosed with uncomplicated cystitis and treated accordingly
- control group: women older than 18 years presented for reasons unlikely to affect the lower urinary tract

SUMMARY:
The goal of this prospective observational study is to provide an Arabic translation of the Acute Cystitis Symptom Score (ACSS) and to test the linguistic validity and clinical reliability of the translated Arabic version of ACCS (Arabic-ACCS) in Arabic-speaking women older than 18 years of age diagnosed with uncomplicated cystitis.

The main questions it aims to answer are:

* Do the questions of the Arabic-ACSS have sufficient clarity?
* Can the Arabic-ACCS serve its purpose in identifying the presence of uncomplicated cystitis in Arabic-speaking women? The participant will be asked to fill out the Arabic-ACCS questionnaire at the time of diagnosis. The participants will be asked to fill out the second part of the Arabic-ACCS questionnaire 5-10 days later after receiving the appropriate treatment according to the local health policy as prescribed by the treating physician.

Researchers will compare the results from the patients who filled out the first part of the questionnaire with the results of a comparable group of women who were presented with complaints unrelated to the lower urinary tract.

ELIGIBILITY:
Inclusion Criteria:

* women.
* presented to the urology or gynecology and obstetrics outpatient clinics.
* having the diagnosis of uncomplicated cystitis.

Exclusion Criteria:

* pregnancy.
* urethral catheterization.
* anatomical abnormality of the urinary tract.
* Neurologic abnormality that affects bladder function.
* urinary tract stones.
* recent antibiotic usage (within 1 month).
* immunosuppression.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women presented to the urology or gynecology and obstetrics outpatient clinics at Alkindy Teaching Hospital and Al-Elwiya Maternity Teaching Hospital having the diagnosis of uncomplicated cystitis will serve as the case group.
  In addition, a control group of women attending the same clinics who are complaining of conditions unlikely to affect the symptoms of the lower urinary tract will be recruited as a control group
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Linguistic validity | 14 days
  Each question in the translated Arabic version of the Acute Cystitis Symptom Score questionnaire should be clear, and the answer to the question should provide the desired piece of information.
  The acute cystitis symptom score questionnaire consists of four domains at the first visit. These domains ask about typical symptoms (6 questions), differential symptoms (4 questions), quality of life (3 questions), and additional information (5 questions). In addition to the aforementioned items, there is a dynamic domain (one question) that is only asked on the second visit.
Clinical reliability | 7 months
  The linguistically validated, translated Arabic version of the Acute Cystitis Symptom Score questionnaire should be able to recognize patients with acceptable specificity and sensitivity.
  The sum of the "typical symptoms," "deferential symptoms," and "quality of life" domain scores can range from 0 to 18, 0 to 12, and 0 to 9, respectively. The lower score signifies less severity; the top score is the most severe grade for each domain.
  The "additional" domain consists of five "yes" or "no" questions designed to discover if there are any criteria that may exclude the diagnosis of uncomplicated cystitis or produce similar symptoms.
  The sum of the "typical symptoms" domain alone will be tested for its diagnostic reliability.
  In addition, the sum of both "typical symptoms" and "quality of life" domains is also to be tested for its diagnostic reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Harth Mohamed Kamber, FICMS (Uro.), Study Chair — University of Baghdad / Alkindy College of Medicine; Zahraa Muhmmed Jameel Al-Sattam, FICMS (Gyn.), Principal Investigator — University of Baghdad / Alkindy College of Medicine; Weqar Akram Hussein, FICMS (Gyn.), Principal Investigator — University of Baghdad / Alkindy College of Medicine; Ahmed Abed Marzook, FICMS, Principal Investigator — Dijlah University College
Locations (2):
- Iraq (2):
  - Al-Elwiya Maternity Teaching Hospital, Baghdad
  - Alkindy Teaching Hospital, Baghdad